CLINICAL TRIAL: NCT00070499
Title: A Phase IIb Study of Molecular Responses to Imatinib, at Standard or Increased Doses, or Dasatinib (BMS-354825) (NSC-732517) for Previously Untreated Patients With Chronic Myelogenous Leukemia (CML) in Chronic Phase
Brief Title: Imatinib Mesylate or Dasatinib in Treating Patients With Previously Untreated Chronic Phase Chronic Myelogenous Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00764; NCI-2009-00764 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S0325; S0325 (Other: SWOG); S0325 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Results first posted 2012-07-10 (Estimated); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Chronic Myeloid Leukemia, BCR-ABL1 Positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (QD imatinib mesylate) (Experimental): Patients receive imatinib mesylate PO QD. Treatment repeats every 4 weeks for up to 5 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Imatinib Mesylate; Other: Laboratory Biomarker Analysis
- Arm II (BID imatinib mesylate) (Experimental): Patients receive imatinib mesylate PO BID. Treatment repeats every 4 weeks for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Imatinib Mesylate; Other: Laboratory Biomarker Analysis
- Arm III (dasatinib) (Experimental): Patients receive dasatinib PO BID. Treatment repeats every 4 weeks for up to 5 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS 354825; BMS-354825; BMS354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
  Arms: Arm III (dasatinib)
Drug: Imatinib Mesylate — Given PO
  Other Names: CGP 57148; CGP 57148B; CGP-57148; CGP-57148B; CGP57148; CGP57148B; Gleevec; Glivec; Imarech; Imat; Imkeldi; STI 571; STI-571; STI571
  Arms: Arm I (QD imatinib mesylate); Arm II (BID imatinib mesylate)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase IIB trial studies imatinib mesylate at two different doses and dasatinib to see how well they work in treating patients with previously untreated chronic phase chronic myelogenous leukemia. Imatinib mesylate or dasatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the molecular response rates, as measured by the decrease in breakpoint cluster region-Abelson murine leukemia viral oncogene homolog 1 (BCR-ABL) transcripts after 12 months of treatment, in patients with previously untreated chronic myelogenous leukemia (CML) in chronic phase who are treated with either dasatinib 100 mg/day or imatinib (STI571, Gleevec) (imatinib mesylate) 400 mg/day.

II. To test whether increasing the dose of imatinib (STI571, Gleevec®) from 400 mg/day to 800 mg/day increases the rate of molecular response, as measured by the decrease in BCR-ABL transcripts after 12 months of treatment, in patients with previously untreated CML in chronic phase.

III. To estimate rates of cytogenetic and hematologic responses to imatinib 400 mg/day, imatinib 800 mg/day, and dasatinib 100 mg/day.

IV. To evaluate in a preliminary manner the prognostic effects of derivative (der)(9) and der(22) chromosomal deletions for response in CML patients treated with imatinib and dasatinib.

V. To investigate in a preliminary manner changes in gene expression at relapse or progression compared to pre-treatment.

VI. To estimate the frequency and severity of toxicities of the three treatment regimens.

VII. To evaluate, in a preliminary manner, the overall survival and relapse-free survival of patients treated with these regimens.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive imatinib mesylate orally (PO) once daily (QD). Treatment repeats every 4 weeks for up to 5 years in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive imatinib mesylate PO twice daily (BID). Treatment repeats every 4 weeks for up to 12 months in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive dasatinib PO BID. Treatment repeats every 4 weeks for up to 5 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have CML in chronic phase based on bone marrow aspiration and biopsy and peripheral blood counts obtained within 28 days before registration
* Patients must be registered on this study within 180 days after the date of first being diagnosed with CML, based on a cytogenetic or molecular analysis of peripheral blood or bone marrow, demonstrating the presence of the Philadelphia chromosome or variants of the (9;22) translocation or testing positive for Bcr-Abl by real time-polymerase chain reaction (RT-PCR); patients may have secondary chromosomal abnormalities in addition to the Philadelphia chromosome and remain eligible
* Patients must have Zubrod performance status 0-2
* Patients must not have received prior treatment for CML with the exception of hydroxyurea and/or anagrelide
* Patients must not have received any prior chemotherapy regimen for peripheral blood stem cell mobilization; (prior collection of unmobilized peripheral blood stem cells is permitted)
* Serum bilirubin =< 2.0 x the institutional upper limit of the normal (IULN)
* Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) or serum glutamate pyruvate transaminase (SGPT)/alanine transaminase (ALT) =< 2.0 x the IULN
* Patients (Southwestern Oncology Group [SWOG] institutions only) must be registered on SWOG-9007, "Cytogenetic Studies in Leukemia Patients;" collection of the pretreatment bone marrow specimen must be completed within 28 days prior to registration; the pretreatment bone marrow specimen must be submitted to an approved Southwest Oncology Group Cytogenetics Laboratory for cytogenetic analysis as described, and an aliquot of the bone marrow (or peripheral blood if the marrow aspiration is a dry tap) must be submitted for fluorescent in situ hybridization (FISH) analysis; note that protocol SWOG-9007 also requires submission of bone marrow specimens at the time of progression to the accelerated or blastic phase of CML or the loss of complete hematologic response and every six months while the patient is on this study
* Patients (SWOG institutions only) must be registered on S9910, "Leukemia Centralized Reference Laboratories and Tissue Repositories, Ancillary;" specimens of peripheral blood and bone marrow must be submitted to the Southwest Oncology Group Lymphoid Leukemia and CML Centralized Laboratory in Seattle, Washington; collection of pretreatment blood and marrow specimens must be completed within 28 days prior to registration; note that this study also requires submission of peripheral blood and bone marrow specimens at various times after entry into the study
* Patients must not have undergone major surgery within 28 days before registration, and must have fully recovered from any other prior major surgery
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, cervical carcinoma in situ, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for five years
* Patients must have an electrocardiogram (ECG) within 42 days prior to registration, and must not have any of the following cardiac symptoms prior to entry on study:

  * Uncontrolled angina, congestive heart failure or myocardial infarction (MI) within 6 months of study entry
  * Diagnosed or suspected congenital long QT syndrome
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
  * Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (> 450 msec)
  * Uncontrolled hypertension
* Patients must not have a history of significant bleeding disorder unrelated to cancer, including:

  * Congenital bleeding disorders (e.g., von Willebrand's disease)
  * Acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and identification (ID) number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2004-08-15 (Actual); Primary Completion 2010-11-01 (Actual); Study Completion 2026-03-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Druker, Principal Investigator — SWOG Cancer Research Network
Locations (341):
- United States (330):
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fremont, Fremont, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - University of Colorado, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Montrose Memorial Hospital, Montrose, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Saint Francis Hospital - Wilmington, Wilmington, Delaware
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Deerpath Medical Associates, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Midwest Cancer Research Group Incorporated, Skokie, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Reid Health, Richmond, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Memorial Hospital of Arkansas City, Arkansas City, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Ottawa, Ottawa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - AdventHealth Shawnee Mission, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - York Hospital, York Village, Maine
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Unspecified Site, Rockville, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Missouri Cancer Associates, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Internal Medicine of Bozeman, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Adirondack Cancer Center, Glens Falls, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Syracuse Veterans Administration Medical Center, Syracuse, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Lenoir Memorial Hospital, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (11):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Verdun Hospital Centre, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Radich JP, Kopecky KJ, Appelbaum FR, Kamel-Reid S, Stock W, Malnassy G, Paietta E, Wadleigh M, Larson RA, Emanuel P, Tallman M, Lipton J, Turner AR, Deininger M, Druker BJ. A randomized trial of dasatinib 100 mg versus imatinib 400 mg in newly diagnosed chronic-phase chronic myeloid leukemia. Blood. 2012 Nov 8;120(19):3898-905. doi: 10.1182/blood-2012-02-410688. Epub 2012 Aug 22. PMID 22915637

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note that 403 patients were registered to the study. Three patients were registered to standard dose imatinib while concurrent randomization was occurring between standard dose imatinib, high dose imatinib, and dasatinib. Those three patients are included in both the standard dose imatinib A and B cohorts.
Groups:
- Standard Dose Imatinib A: Randomization between occurred between standard dose imatinib A and high dose imatinib. Standard dose imatinib was 400 mg daily.
- High Dose Imatinib: High dose imatinib was 800 mg daily.
- Dasatinib: Dasatinib dose was 100 mg daily
- Standard Dose Imatinib B: Randomization occurred between Standard dose imatinib and dasatinib. Standard dose imatinib was 400 mg daily.
Period: Overall Study
Arm/Group | Standard Dose Imatinib A | High Dose Imatinib | Dasatinib | Standard Dose Imatinib B
Started | 75 | 78 | 126 | 127
Eligible | 73 | 73 | 123 | 125
Eligible and Treated | 72 | 73 | 123 | 123
Completed | 37 | 52 | 6 | 17
Not Completed | 38 | 26 | 120 | 110
Not completed — Adverse Event | 6 | 6 | 19 | 15
Not completed — Refusal unrelated to adverse effects | 7 | 5 | 5 | 8
Not completed — Progression/relapse | 4 | 2 | 1 | 4
Not completed — Death | 1 | 1 | 1 | 2
Not completed — Other - not protocol specified | 7 | 3 | 12 | 20
Not completed — Still on protocol treatment | 10 | 4 | 79 | 57
Not completed — Did not start treatment | 1 | 0 | 0 | 2
Not completed — Not eligible | 2 | 5 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Standard Dose Imatinib A: Randomization between occurred between standard dose imatinib A and high dose imatinib
- Standard Dose Imatinib B: Randomization occurred between Standard dose imatinib and dasatinib
- Total: Total of all reporting groups
Arm/Group | Standard Dose Imatinib A | High Dose Imatinib | Dasatinib | Standard Dose Imatinib B | Total
Number analyzed (Participants) | 72 | 73 | 123 | 123 | 391
Age, Continuous [Median (Full Range); unit: years] | 50 [23 to 80] | 52 [20 to 82] | 47 [18 to 90] | 50 [19 to 89] | 50 [18 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 48 | 51 | 151
  Male | 46 | 47 | 75 | 72 | 240
Region of Enrollment [Number; unit: participants]
  United States | 72 | 73 | 123 | 123 | 391

OUTCOME MEASURES:

1. Primary Outcome: Molecular Response Rate at 12 Months
Description: Median value of baseline bcr-abl/bcr ratio from pretreatment was used as the baseline value for assessing each patient's molecular response. Molecular response criteria were: 1) not failed treatment on or before 12-month evaluation; 2) met criteria for hemalotogic response; 3) bcr-abl/bcr ration at 12-months must be 10,000 times smaller than the pretreatment ratio.
Time Frame: pretreatment and after 12 months of treatment
Population: Patients with follow-up specimens assayed by reverse transcription polymerase chain reaction (RT-PCR)
Measure: Number; unit: participants
Groups:
- Standard Dose Imatinib A: Standard dose imatinib A
- High Dose Imatinib: High dose imatinib
- Dasatinib: Dasatinib
- Standard Dose Imatinib B: Standard dose imatinib B
Arm/Group | Standard Dose Imatinib A | High Dose Imatinib | Dasatinib | Standard Dose Imatinib B
Number analyzed (Participants) | 49 | 55 | 99 | 90
participants | 5 | 14 | 27 | 18
Statistical Analysis 1: Comparison: Standard Dose Imatinib A vs High Dose Imatinib; Test type: Superiority or Other; p = 0.073, Fisher Exact
Statistical Analysis 2: Comparison: Dasatinib vs Standard Dose Imatinib B; Test type: Superiority or Other; p = 0.31, Fisher Exact

2. Secondary Outcome: Hematologic Response
Description: Hematologic response assesses whether patients' blood counts return to normal
Time Frame: 1 month after starting treatment
Population: Eligible, treated patients who were evaluable for hematologic response
Measure: Number; unit: participants
Arm/Group | Standard Dose Imatinib A | High Dose Imatinib | Dasatinib | Standard Dose Imatinib B
Number analyzed (Participants) | 72 | 72 | 123 | 123
participants | 63 | 66 | 107 | 112

3. Secondary Outcome: 2-year Overall Survival (OS)
Description: Overall survival was measured from the date of registration to study until death from any cause with observations censored at the date of last contact for patients last known to be alive.
Time Frame: Every three months for the first year, every six months in years 2 and 3, and annually for years 4 and 5
Population: All eligible patients who were treated
Measure: Number; unit: Percent of population
Arm/Group | Standard Dose Imatinib A | High Dose Imatinib | Dasatinib | Standard Dose Imatinib B
Number analyzed (Participants) | 72 | 73 | 123 | 123
Percent of population | 89 | 95 | 97 | 98
Statistical Analysis 1: Comparison: Standard Dose Imatinib A vs High Dose Imatinib; Log-rank test of overall survival; Test type: Superiority or Other; p = 0.29, Log Rank
Statistical Analysis 2: Comparison: Dasatinib vs Standard Dose Imatinib B; Log-rank test of overall survival; Test type: Superiority or Other; p = 0.55, Log Rank

4. Secondary Outcome: Two Year Relapse-free Survival
Description: Relapse-free survival is measured from the date of documented (possibly unconfirmed) hematologic complete remission until loss of hematologic complete remission or death from any cause. Observations are censored at the date of last contact for patients last known to be alive with report of loss of hematologic complete remission.
Time Frame: every 3 months for the first year, every six months for years 2 and 3, annually for years 4 and 5
Population: Eligible, treated patients who achieved a hematologic complete remission
Measure: Number; unit: Percent of population
Arm/Group | Standard Dose Imatinib A | High Dose Imatinib | Dasatinib | Standard Dose Imatinib B
Number analyzed (Participants) | 63 | 66 | 107 | 112
Percent of population | 83 | 97 | 96 | 95
Statistical Analysis 1: Comparison: Standard Dose Imatinib A vs High Dose Imatinib; Log-rank test of relapse-free survival; Test type: Superiority or Other; p = 0.074, Log Rank
Statistical Analysis 2: Comparison: Dasatinib vs Standard Dose Imatinib B; Log-rank test of relapse-free survival; Test type: Superiority or Other; p = 0.29, Log Rank

5. Secondary Outcome: Toxicity
Description: Number of patients with Grade 3-5 adverse events that are related to study drug by given type of adverse event
Time Frame: Patients were assessed for adverse events monthly every 4 weeks for the first year, every 6 months for years 2 and 3, and annually for years 4 and 5.
Population: Eligible patients who started therapy
Measure: Number; unit: Participants with a given type of AE
Groups:
- Standard Dose Imatinib A: Randomization occurred between standard dose imatinib A and high dose imatinib. patients received 400 mg imatinib daily
- High Dose Imatinib: Patients received 800 mg imatinib daily
- Dasatinib: Patients received 100 mg dasatinib daily
- Standard Dose Imatinib B: Randomization occurred between Standard dose imatinib B and dasatinib. patients received 400 mg imatinib daily
Arm/Group | Standard Dose Imatinib A | High Dose Imatinib | Dasatinib | Standard Dose Imatinib B
Number analyzed (Participants) | 72 | 72 | 122 | 123
Participants with a given type of AE
  ALT, SGPT (serum glutamic pyruvic transaminase) | 1 | 3 | 1 | 3
  AST, SGOT (serum glutamic oxaloacetic trans.) | 1 | 1 | 1 | 2
  Bilirubin (hyperbilirubinemia) | 1 | 0 | 0 | 0
  Bronchospasm, wheezing | 0 | 0 | 0 | 1
  CNS cerebrovascular ischemia | 0 | 0 | 1 | 0
  CPK (creatine phosphokinase) | 3 | 0 | 1 | 0
  Cardiac-ischemia/infarction | 0 | 0 | 2 | 0
  Colitis | 0 | 0 | 3 | 0
  Conduction abnor/Atrioventricular heart block | 0 | 0 | 1 | 0
  Constipation | 0 | 0 | 1 | 0
  Dehydration | 0 | 0 | 1 | 0
  Diarrhea | 1 | 6 | 6 | 2
  Distention/bloating, abdominal | 0 | 1 | 0 | 0
  Dizziness | 1 | 0 | 0 | 1
  Dyspnea (shortness of breath) | 0 | 2 | 7 | 2
  Edema: head and neck | 2 | 0 | 0 | 2
  Edema: limb | 0 | 2 | 1 | 1
  Edema: trunk/genital | 0 | 1 | 0 | 0
  Edema: viscera | 1 | 0 | 0 | 0
  Fatigue (asthenia, lethargy, malaise) | 0 | 11 | 1 | 1
  Febrile neutropenia | 1 | 1 | 3 | 0
  GGT (gamma-glutamyl transpeptidase) | 0 | 1 | 0 | 0
  Glucose, serum-high (hyperglycemia) | 0 | 0 | 3 | 0
  Hematoma | 0 | 0 | 1 | 0
  Hemoglobin | 5 | 8 | 12 | 5
  Hepatobiliary/Pancreas-Other (Specify) | 0 | 1 | 0 | 0
  Hot flashes/flushes | 0 | 0 | 1 | 0
  Hypertension | 0 | 0 | 1 | 0
  Hypoxia | 0 | 1 | 0 | 0
  Infection with Grade 3 or 4 neutrophils - Blood | 0 | 0 | 1 | 0
  Infection with Grade 3/4 neut - Lung (pneumon | 0 | 0 | 2 | 0
  Infec with norm ANC or Grade 1 or 2 neut - Colon | 0 | 1 | 0 | 0
  Inf with no ANC or Grade 1/2 netLung (pneumonia) | 0 | 1 | 2 | 0
  Infec with norm ANC or Grade 1 or 2 neut - Scrotum | 0 | 0 | 1 | 0
  Infect with norm ANC or Grade 1 or 2 neut - Sinus | 0 | 0 | 1 | 0
  Inf with no ANC or Grade 1/2 neut - Ur tract NOS | 1 | 0 | 0 | 0
  Infection with unknown ANC - Sinus | 0 | 0 | 1 | 0
  Left ventricular diastolic dysfunction | 0 | 0 | 1 | 0
  Leukocytes (total WBC) | 1 | 2 | 3 | 3
  Lymphopenia | 1 | 1 | 3 | 1
  Metabolic/Laboratory-Other (Specify) | 0 | 0 | 1 | 0
  Mood alteration - depression | 1 | 0 | 0 | 0
  Mucositis/stomatitis (clinical exam) - Oral cavity | 0 | 0 | 0 | 2
  Muscle weak, not due to neurop. Whole body/general | 0 | 1 | 0 | 0
  Nausea | 2 | 2 | 0 | 1
  Neuropathy: motor | 0 | 0 | 1 | 0
  Neuropathy: sensory | 0 | 0 | 1 | 0
  Neutrophils/granulocytes (ANC/AGC) | 8 | 12 | 18 | 15
  Pain - Abdomen NOS | 1 | 4 | 3 | 1
  Pain - Back | 0 | 1 | 0 | 1
  Pain - Bone | 1 | 3 | 2 | 0
  Pain - Chest/thorax NOS | 0 | 1 | 1 | 1
  Pain - Extremity-limb | 0 | 1 | 0 | 0
  Pain - Head/headache | 1 | 1 | 3 | 3
  Pain - Joint | 0 | 1 | 1 | 2
  Pain - Muscle | 1 | 3 | 0 | 1
  Pain-Other (Specify) | 0 | 0 | 0 | 1
  Pericardial effusion (non-malignant) | 0 | 0 | 3 | 0
  Phosphate, serum-low (hypophosphatemia) | 0 | 0 | 1 | 1
  Platelets | 6 | 14 | 22 | 11
  Pleural effusion (non-malignant) | 0 | 0 | 4 | 1
  Potassium, serum-high (hyperkalemia) | 0 | 0 | 1 | 0
  Potassium, serum-low (hypokalemia) | 0 | 0 | 1 | 2
  Prolonged QTc interval | 0 | 0 | 1 | 0
  Proteinuria | 0 | 0 | 1 | 0
  Pruritus/itching | 0 | 1 | 0 | 2
  Pulmonary/Upper Respiratory-Other (Specify) | 0 | 0 | 1 | 0
  Rash/desquamation | 1 | 4 | 0 | 2
  Rash: acne/acneiform | 0 | 0 | 1 | 0
  Restrictive cardiomyopathy | 0 | 1 | 0 | 0
  Retinal detachment | 0 | 0 | 0 | 1
  Sodium, serum-high (hypernatremia) | 0 | 0 | 1 | 0
  Syncope (fainting) | 0 | 0 | 1 | 0
  Vaginal mucositis | 0 | 0 | 1 | 0
  Vision-blurred vision | 1 | 1 | 1 | 0
  Vomiting | 1 | 0 | 1 | 0
  Watery eye (epiphora, tearing) | 0 | 0 | 1 | 0
  Weight gain | 0 | 1 | 3 | 0

ADVERSE EVENTS:
Time Frame: While the patient is on treatment until resolution of acute toxicities with maximum grade reported
Description: Regular investigator assessments are reported after each cycle of protocol treatment
Groups:
- Standard Dose Imatinib A: Randomization occurred between standard dose imatinib A and high dose imatinib/ patients received 400 mg imatinib daily
- Standard Dose Imatinib B: Randomization occurred between Standard dose imatinib B and dasatinib/ patients received 400 mg imatinib daily
Arm/Group | Standard Dose Imatinib A | High Dose Imatinib | Dasatinib | Standard Dose Imatinib B
Serious Adverse Events (participants affected / at risk) | 4/72 | 0/72 | 20/122 | 0/123
Other Adverse Events (participants affected / at risk) | 71/72 | 72/72 | 115/122 | 120/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose Imatinib A (N=72) | High Dose Imatinib (N=72) | Dasatinib (N=122) | Standard Dose Imatinib B (N=123)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (non-malignant) (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ulcer, GI - Duodenum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema: limb (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain - Chest/thorax NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Lung (pneumon (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Scrotum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Sinus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CPK (creatine phosphokinase) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelets (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prolonged QTc interval (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain - Head/headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood alteration - depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose Imatinib A (N=72) | High Dose Imatinib (N=72) | Dasatinib (N=122) | Standard Dose Imatinib B (N=123)
Hemoglobin (Blood and lymphatic system disorders) | 47 (47) | 59 (59) | 86 (86) | 87 (87)
Vision-blurred vision (Eye disorders) | 5 (5) | 4 (4) | 0 (0) | 7 (7)
Watery eye (epiphora, tearing) (Eye disorders) | 0 (0) | 10 (10) | 0 (0) | 13 (13)
Ascites (non-malignant) (Gastrointestinal disorders) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 6 (6) | 9 (9) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 26 (26) | 40 (40) | 41 (41) | 51 (51)
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Flatulence (Gastrointestinal disorders) | 0 (0) | 9 (9) | 11 (11) | 9 (9)
Heartburn/dyspepsia (Gastrointestinal disorders) | 7 (7) | 19 (19) | 12 (12) | 22 (22)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 36 (36) | 42 (42) | 33 (33) | 63 (63)
Pain - Abdomen NOS (Gastrointestinal disorders) | 7 (7) | 19 (19) | 16 (16) | 16 (16)
Vomiting (Gastrointestinal disorders) | 11 (11) | 19 (19) | 19 (19) | 25 (25)
Edema: head and neck (General disorders) | 28 (28) | 43 (43) | 14 (14) | 45 (45)
Edema: limb (General disorders) | 26 (26) | 29 (29) | 21 (21) | 36 (36)
Edema: trunk/genital (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 47 (47) | 57 (57) | 66 (66) | 67 (67)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC lt1.0 x 10e9/L) (General disorders) | 4 (4) | 9 (9) | 15 (15) | 7 (7)
Pain - Chest/thorax NOS (General disorders) | 0 (0) | 7 (7) | 11 (11) | 0 (0)
Rigors/chills (General disorders) | 4 (4) | 5 (5) | 0 (0) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 6 (6) | 12 (12) | 20 (20) | 15 (15)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 9 (9) | 18 (18) | 23 (23) | 18 (18)
Alkaline phosphatase (Investigations) | 14 (14) | 23 (23) | 20 (20) | 26 (26)
Bilirubin (hyperbilirubinemia) (Investigations) | 5 (5) | 11 (11) | 7 (7) | 0 (0)
Creatinine (Investigations) | 10 (10) | 12 (12) | 13 (13) | 18 (18)
Leukocytes (total WBC) (Investigations) | 14 (14) | 28 (28) | 34 (34) | 35 (35)
Lymphopenia (Investigations) | 8 (8) | 8 (8) | 10 (10) | 8 (8)
Metabolic/Laboratory-Other (Specify) (Investigations) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 22 (22) | 33 (33) | 46 (46) | 45 (45)
Platelets (Investigations) | 23 (23) | 46 (46) | 71 (71) | 42 (42)
Prolonged QTc interval (Investigations) | 0 (0) | 7 (7) | 0 (0) | 0 (0)
Weight gain (Investigations) | 6 (6) | 17 (17) | 18 (18) | 17 (17)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 (5) | 12 (12) | 9 (9) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 11 (11) | 16 (16) | 22 (22) | 12 (12)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 (4) | 10 (10) | 12 (12) | 10 (10)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 10 (10) | 11 (11) | 15 (15) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5 (5) | 4 (4) | 9 (9) | 9 (9)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 0 (0) | 7 (7)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 9 (9) | 11 (11) | 9 (9) | 8 (8)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 11 (11) | 15 (15) | 26 (26) | 21 (21)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 22 (22) | 29 (29) | 15 (15) | 47 (47)
Dizziness (Nervous system disorders) | 4 (4) | 9 (9) | 13 (13) | 10 (10)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 0 (0) | 15 (15) | 0 (0)
Pain - Head/headache (Nervous system disorders) | 9 (9) | 9 (9) | 33 (33) | 23 (23)
Taste alteration (dysgeusia) (Nervous system disorders) | 0 (0) | 9 (9) | 0 (0) | 8 (8)
Insomnia (Psychiatric disorders) | 8 (8) | 10 (10) | 0 (0) | 11 (11)
Mood alteration - depression (Psychiatric disorders) | 5 (5) | 6 (6) | 8 (8) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 9 (9) | 7 (7)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6) | 22 (22) | 12 (12)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 7 (7) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 16 (16) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6) | 11 (11) | 10 (10)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6 (6) | 20 (20) | 11 (11) | 18 (18)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 19 (19) | 36 (36) | 41 (41) | 35 (35)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 12 (12) | 0 (0)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 5 (5) | 10 (10) | 8 (8) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less